CLINICAL TRIAL: NCT06490302
Title: Clinical Evaluation of Biomedics Monthly Toric and Avaira Vitality Toric
Brief Title: Clinical Evaluation of Two Toric Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-157
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens A (ocufilcon D) (Experimental): All participants will wear lens A for 15 minutes (Period 1).
  Interventions: Device: Lens A (ocufilcon D)
- Lens B (fanfilcon A) (Experimental): All participants will wear lens B for 15 minutes (Period 2).
  Interventions: Device: Lens B (fanfilcon A)

INTERVENTIONS:
Device: Lens A (ocufilcon D) — 15 minutes of daily wear
  Arms: Lens A (ocufilcon D)
Device: Lens B (fanfilcon A) — 15 minutes of daily wear
  Arms: Lens B (fanfilcon A)

SUMMARY:
The aim of this study is to compare the short-term clinical performance of two toric contact lenses.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the short-term clinical performance of two toric contact lenses when compared to each other after 15 minutes of daily wear each.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 40 years of age (inclusive)
* Has had a self-reported visual exam in the last two years.
* Is an adapted soft contact lens wearer.
* Is not a habitual wearer of either study lens.
* Has a contact lens spherical prescription between +5.00 to -9.00 (inclusive) best corrected visual acuity of 20/30 or better in either eye.
* Have contact lens prescription of no less than -0.75D of astigmatism and no more than -2.25D in both eyes.
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease.
* Has read, understood and signed the informed consent letter.
* Patient contact lens refraction should fit within the available parameters of the study lenses.
* Is willing to comply with the wear schedule (at least 5 days per week, >8 hours/day assuming there are no contraindications for doing so).
* Is willing to comply with the visit schedule.

Exclusion Criteria:

* Has a CL prescription outside the range of the available parameters of the study lenses.
* Has a spectacle cylinder less than -0.75D or more than -2.50D of cylinder in either eye.
* Slit lamp findings that would contraindicate contact lens wear such as:

  1. Pathological dry eye or associated findings
  2. Pterygium, pinguecula, or corneal scars within the visual axis
  3. Neovascularization > 0.75 mm in form of the limbus
  4. Giant papillary conjuctivitis (GCP) worse than grade 1
  5. Anterior uveitis or iritis (past or present)
  6. Seborrheic eczema, seborrheic conjunctivitis
  7. History of corneal ulcers or fungal infections
  8. Poor personal hygiene
  9. Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
  10. Has aphakia, keratoconus or a highly irregular cornea.
  11. Has Presbyopia or has dependence on spectacles for near work over the contact lenses.
  12. Has undergone corneal refractive surgery.
  13. Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Guerrero, MSc, FIACLE, Principal Investigator — National Autonomous University
Locations (1):
- Consultorio Optométrico Queretaro, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty participants were screened. All the participants who were eligible in the study were included in the analysis. (n=40)
Groups:
- Lens A (Ocufilcon D): All participants wore lens A for 15 minutes (Period 1).
  Lens A (ocufilcon D): 15 minutes of daily wear
- Lens B (Fanfilcon A): All participants wore lens B for 15 minutes (Period 2).
  Lens B (fanfilcon A): 15 minutes of daily wear
Period: Period 1: Lens A (15 Minutes)
Arm/Group | Lens A (Ocufilcon D) | Lens B (Fanfilcon A)
Started | 40 | 0 (All participants received Lens A in Period 1.)
Completed | 40 | 0
Not Completed | 0 | 0
Period: Period 2: Lens B (15 Minutes)
Arm/Group | Lens A (Ocufilcon D) | Lens B (Fanfilcon A)
Started | 0 (All participants received Lens B in Period 2.) | 40
Completed | 0 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Includes all Study Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.6 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall Fit Acceptance
Description: Overall lens fit acceptance was measured on a scale from 0-4 (0= Should not be worn, 4= Perfect)
Time Frame: At the end of 15 minutes of daily wear
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lens A (Ocufilcon D) | Lens B (Fanfilcon A)
Number analyzed (Participants) | 40 | 40
units on a scale | 3.6 (0.8) | 3.7 (0.6)

ADVERSE EVENTS:
Time Frame: Duration of the study, approximately 4 weeks.
Arm/Group | Lens A (Ocufilcon D) | Lens B (Fanfilcon A)
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT06490302/Prot_SAP_000.pdf